CLINICAL TRIAL: NCT03769181
Title: A Phase 1/2 Open-label, Multi-center, Safety, Preliminary Efficacy and Pharmacokinetic (PK) Study of Isatuximab in Combination With Other Anti-cancer Therapies in Participants With Lymphoma
Brief Title: A Study of Isatuximab-based Therapy in Participants With Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was stopped after interim analysis for all 4 cohorts with results either not fulfilling the pre-planned interim analysis criteria or fulfilling the criteria but as per sponsor decision. It was not due to any safety concern
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT15320; 2018-002442-37 (EudraCT Number); U1111-1211-9010 (Registry Identifier: ICTRP)
Record Dates: First submitted 2018-11-29; First posted 2018-12-07 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Lymphoma | interventions — isatuximab; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort A1: cHL: Isatuximab + Cemiplimab (Experimental): Classic Hodgkin's lymphoma (cHL), anti-programmed cell death protein 1/ligand 1 (PD-1/PD-L1) inhibitor naïve participants received isatuximab 10 milligrams per kilogram (mg/kg), intravenous (IV) infusion once a week (QW) in Cycle 1 and then every 2 weeks (Q2W) from Cycle 2 to Cycle 6 (each cycle of 28 days), and then every 3 weeks (Q3W) from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 milligrams (mg) Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, with optional radiotherapy until, unacceptable adverse events (AEs) or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of complete response [CR], whichever was longer) of delivery of investigational medicinal product(s) without documented progressive disease (PD), or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
  Interventions: Drug: isatuximab SAR650984; Drug: cemiplimab REGN2810
- Cohort A2: cHL: Isatuximab + Cemiplimab (Experimental): cHL, anti-PD-1/PD-L1 inhibitor progressor participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, with optional radiotherapy until, unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
  Interventions: Drug: isatuximab SAR650984; Drug: cemiplimab REGN2810
- Cohort B: DLBCL: Isatuximab + Cemiplimab (Experimental): Diffuse large B-cell lymphoma (DLBCL), anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30 until, unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
  Interventions: Drug: isatuximab SAR650984; Drug: cemiplimab REGN2810
- Cohort C: PTCL: Isatuximab + Cemiplimab (Experimental): Peripheral T-cell lymphoma (PTCL), anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30 until, unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
  Interventions: Drug: isatuximab SAR650984; Drug: cemiplimab REGN2810

INTERVENTIONS:
Drug: isatuximab SAR650984 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Sarclisa
Drug: cemiplimab REGN2810 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous

SUMMARY:
Primary Objectives:

Phase 1

-To characterize the safety and tolerability of isatuximab in combination with cemiplimab in participants with relapsed and refractory classic Hodgkin's lymphoma (cHL), diffuse large B-cell lymphoma (DLBCL) or peripheral T-cell lymphoma (PTCL), and to confirm the recommended Phase 2 dose (RP2D).

Phase 2

* Cohort A1 (anti-programmed cell death protein 1/ligand 1 [PD-1/PD-L1] naïve cHL): To assess the complete remission (CR) rate of isatuximab in combination with cemiplimab.
* Cohort A2 (cHL progressing from PD-1/PD-L1), B (DLBCL) and C (PTCL): To assess the objective response rate (ORR) of isatuximab in combination with cemiplimab.

Secondary Objectives:

* To evaluate the safety of the RP2D of the combination of isatuximab with cemiplimab.
* To evaluate the safety of the combination of isatuximab with cemiplimab and radiotherapy in participants with cHL.
* To evaluate the immunogenicity of isatuximab and cemiplimab when given in combination.
* To characterize the pharmacokinetic (PK) profile of isatuximab and cemiplimab when given in combination.
* To assess overall efficacy of isatuximab in combination with cemiplimab and isatuximab in combination with cemiplimab and radiotherapy.

DETAILED DESCRIPTION:
The total study duration per participant was up to 28 months, including an up to 28-day screening period, an up to 96-week treatment period, and a 90-day safety follow up period.

ELIGIBILITY:
Inclusion criteria:

* Participants greater than or equal to (>=) 12 years of age inclusive, at the time of signing the informed consent.
* Disease location amenable to tumor biopsy at Baseline.
* Measurable disease.
* For Cohort A1 (cHL anti-programmed cell death protein 1/ligand 1 [PD-1/PD-L1] inhibitor naïve): Histologically confirmed advanced cHL that had relapsed or progressed after at least 3 lines of systemic therapy that included autologous hematopoietic stem cell transplant (auto-HSCT) or auto-HSCT and brentuximab vedotin (BV).
* For Cohort A2 (cHL anti-PD-1/PD-L1 inhibitor progressor): Histologically confirmed advanced cHL which had relapsed or progressed after one previous anti-PD-1/PD-L1 containing regimen as the most recent prior therapy but no more than 4 lines of previous chemotherapy including the anti-PD-1/PD-L1 containing regimen and documentation of benefit during or after the anti-PD-1/PD-L1 containing regimen within 4 months prior to initiation of investigational medicinal product.
* For Cohort B (diffuse large B-cell lymphoma [DLBCL]): Histologically confirmed advanced DLBCL that had relapsed or progressed after 2 lines of systemic therapy including auto-HSCT or 2 lines of systemic therapy for participants who were not eligible for auto-HSCT.
* For Cohort C (peripheral T-cell lymphoma [PTCL]): Histologically confirmed advanced PTCL that had relapsed or progressed after either first-line chemotherapy and auto-HSCT as consolidation of first remission or first-line chemotherapy if participants were ineligible for auto-HSCT.
* Body weight of greater than (>) 45 kilograms for participants with age less than (<)18 years.

Exclusion criteria:

* Prior exposure to agent that blocks CD38.
* For participants with cHL (PD-1/PD-L1 naïve), DLBCL or PTCL prior exposure to any agent (approved or investigational) that blocks the PD-1/PD-L1, PD-L2, CD137, cytotic T-lymphocyte-associated protein 4 or LAG-3.
* Evidence of other immune related disease/conditions.
* Had received a live-virus vaccination within 28 days of planned treatment start; seasonal flu vaccines that do not contain live virus are permitted.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) >=2.
* Poor bone marrow reserve.
* Poor organ function.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (20):
- France (5):
  - Investigational Site Number :2500005, Dijon
  - Investigational Site Number :2500004, Montpellier
  - Investigational Site Number :2500002, Nantes
  - Investigational Site Number :2500007, Pessac
  - Investigational Site Number :2500001, Villejuif
- Italy (3):
  - Investigational Site Number :3800003, Rozzano, Milano
  - Investigational Site Number :3800002, Bologna
  - Investigational Site Number :3800006, Brescia
- Netherlands (2):
  - Investigational Site Number :5280002, Amsterdam
  - Investigational Site Number :5280001, Maastricht
- Portugal (3):
  - Investigational Site Number :6200002, Coimbra
  - Investigational Site Number :6200004, Lisbon
  - Investigational Site Number :6200003, Porto
- South Korea (2):
  - Investigational Site Number :4100001, Gangnam-gu, Seoul-teukbyeolsi
  - Investigational Site Number :4100002, Seoul, Seoul-teukbyeolsi
- Spain (4):
  - Investigational Site Number :7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240005, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number :7240002, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number :7240004, Madrid / Madrid, Madrid, Comunidad de
- Investigational Site Number :1580002, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Carlo-Stella C, Zinzani PL, Sureda A, Araujo L, Casasnovas O, Carpio C, Yeh SP, Bouabdallah K, Cartron G, Kim WS, Cordoba R, Koh Y, Re A, Alves D, Chamuleau M, Le Gouill S, Lopez-Guillermo A, Moreira I, van der Poel MWM, Abbadessa G, Meng R, Ji R, Lepine L, Saleem R, Ribrag V. A phase 1/2, open-label, multicenter study of isatuximab in combination with cemiplimab in patients with lymphoma. Hematol Oncol. 2023 Feb;41(1):108-119. doi: 10.1002/hon.3089. Epub 2022 Oct 31. PMID 36251503
- See also: ACT15320 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25185&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 20 sites in 7 countries. A total of 58 participants were enrolled between 11 December 2018 and 27 August 2020 and received isatuximab in combination with cemiplimab. Study was planned to be conducted in 2 parts: Phase 1(safety run-in) and Phase 2 (efficacy/2-stage design).
Pre-assignment Details: Efficacy results observed in Cohorts B & C didn't fulfill preplanned interim analysis criteria allowing the study to move to Phase(Ph) 2 Stage 2 in these cohorts. Efficacy results observed in Cohorts A1 & A2 fulfilled preplanned interim analysis criteria in Stage 1 to move to Ph 2 Stage 2 in these cohorts. However, study was stopped for all cohorts per sponsor's decision. Participant flow, Baseline,outcome measures & safety data were prespecified to be analyzed on combined Ph 1 & 2 populations.
Groups:
- Cohort A1: cHL: Isatuximab + Cemiplimab: Classic Hodgkin's lymphoma (cHL), anti-programmed cell death protein 1/ligand 1 (PD-1/PD-L1) inhibitor naïve participants with received isatuximab 10 mg/kg, IV infusion once a week (QW) in Cycle 1 and then every 2 weeks (Q2W) from Cycle 2 to Cycle 6 (each cycle of 28 days), and then every 3 weeks (Q3W) from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, with optional radiotherapy until unacceptable adverse events (AEs) or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of complete response [CR], whichever was longer) of delivery of investigational medicinal product(s) without documented progressive disease (PD), or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort A2: cHL: Isatuximab + Cemiplimab: cHL, anti-PD-1/PD-L1 inhibitor progressor participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, with optional radiotherapy until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort B: DLBCL: Isatuximab + Cemiplimab: Diffuse large B-cell lymphoma (DLBCL), anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort C: PTCL: Isatuximab + Cemiplimab: Peripheral T-cell lymphoma (PTCL), anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Period: Overall Study
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Started | 18 | 12 | 17 | 11
Completed (Participants who completed study treatment.) | 5 | 4 | 0 | 0
Not Completed | 13 | 8 | 17 | 11
Not completed — Adverse Event | 1 | 0 | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1
Not completed — Progressive disease | 9 | 7 | 13 | 6
Not completed — Other - Unspecified | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all treated population which included all participants who signed the study informed consent and received at least 1 dose of the study treatment, either isatuximab or cemiplimab.
Groups:
- Cohort A1: cHL: Isatuximab + Cemiplimab: cHL, PD-1/PD-L1 inhibitor naïve participants received isatuximab 10 mg/kg, IV infusion QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days), and then Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, with optional radiotherapy until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort B: DLBCL: Isatuximab + Cemiplimab: DLBCL, anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort C: PTCL: Isatuximab + Cemiplimab: PTCL, anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Total: Total of all reporting groups
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab | Total
Number analyzed (Participants) | 18 | 12 | 17 | 11 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (20.1) | 38.0 (15.5) | 60.8 (14.2) | 65.5 (8.8) | 52.0 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 5 | 4 | 22
  Male | 10 | 7 | 12 | 7 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 4 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 12 | 4 | 8 | 7 | 31
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 5 | 2 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs: Adverse Events (AEs) occurring during 1st treatment cycle, unless due to disease progression or obviously unrelated cause which included: hematological abnormalities: Grade(G) 4 neutropenia(N) for 7 or more consecutive days, G3 to G4 N with fever (temperature greater than or equal to [>=] 38.5 degree Celsius on more than 1 occasion) or microbiologically/radiographically documented infection, G3 to G4 thrombocytopenia with clinically significant bleeding requiring clinical intervention or non-hematological abnormalities: G 4 non-hematologic AE, G>=2 uveitis, G3 non-hematological AE lasting greater than (>)3 days, delay in initiation of Cycle 2 >14 days due to treatment related laboratory abnormalities/AE. Any other AE that the study committee deemed to be dose-limiting, regardless of grade, was also considered as DLT.
Time Frame: Cycle 1 (28 days)
Population: Analysis was performed on DLT evaluable population which included all participants who received the planned doses of isatuximab and cemiplimab during Cycle 1 and completed the DLT observation period after the first administration of the study drug. Here, "0" in the "overall number of participants analyzed" signifies that no participants were evaluable for DLTs in the Cohort A1 arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 0 | 1 | 3 | 1
Participants |  | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. Serious adverse events (SAEs) were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed, worsened or became serious during the TEAE period (defined as the time from the first dose of study treatment up to 30 days after the last dose of study treatment).
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: up to 103 weeks)
Population: Analysis was performed on all treated population which included all participants who signed the informed consent and received at least 1 dose of the study treatment, either isatuximab or cemiplimab.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort C: PTCL: Isatuximab + Cemiplimab: PTCL, anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 12 | 17 | 11
Participants
  TEAEs | 16 | 12 | 17 | 11
  TESAEs | 3 | 2 | 10 | 7

3. Primary Outcome: Number of Participants With Laboratory Abnormalities: Hematological Parameters
Description: Hematological parameters assessed were anemia, white blood cell (WBC) decreased, platelet count decreased, lymphocyte count decreased, and neutrophil count decreased. Abnormality criteria was assessed as per the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 NCI-CTCAE v 5.0), where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: up to 103 weeks)
Population: Analysis was performed on all treated population.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B: DLBCL: Isatuximab + Cemiplimab: DLBCL, anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion Q2W Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 12 | 17 | 11
Participants
  Anemia: Grade 1 | 9 | 6 | 7 | 6
  Anemia: Grade 2 | 5 | 1 | 7 | 3
  Anemia: Grade 3 | 2 | 0 | 2 | 2
  Anemia: Grade 4 | 0 | 0 | 0 | 0
  White blood cell decreased: Grade 1 | 10 | 2 | 9 | 3
  White blood cell decreased: Grade 2 | 1 | 1 | 2 | 4
  White blood cell decreased: Grade 3 | 0 | 0 | 1 | 2
  White blood cell decreased: Grade 4 | 0 | 0 | 2 | 0
  Platelet count decreased: Grade 1 | 8 | 3 | 7 | 3
  Platelet count decreased: Grade 2 | 0 | 0 | 2 | 1
  Platelet count decreased: Grade 3 | 0 | 0 | 0 | 1
  Platelet count decreased: Grade 4 | 0 | 0 | 2 | 3
  Lymphocyte count decreased: Grade 1 | 4 | 2 | 2 | 0
  Lymphocyte count decreased: Grade 2 | 3 | 0 | 4 | 6
  Lymphocyte count decreased: Grade 3 | 5 | 1 | 6 | 3
  Lymphocyte count decreased: Grade 4 | 1 | 0 | 2 | 1
  Neutrophil count decreased: Grade 1 | 0 | 0 | 2 | 2
  Neutrophil count decreased: Grade 2 | 3 | 0 | 2 | 2
  Neutrophil count decreased: Grade 3 | 0 | 0 | 1 | 1
  Neutrophil count decreased: Grade 4 | 0 | 0 | 2 | 2

4. Primary Outcome: Number of Participants With Laboratory Abnormalities: Electrolytes
Description: Electrolyte parameters assessed were hyponatremia, hypokalemia, hyperkalemia, hypocalcemia, hypercalcemia, hypoalbuminemia, hypoglycemia and hyperglycemia. Abnormal criteria was assessed as per the NCI-CTCAE v 5.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: up to 103 weeks)
Population: Analysis was performed on all treated population. Here "number analyzed" signifies the participants with available data for each specified parameter.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A1: cHL: Isatuximab + Cemiplimab: cHL, PD-1/PD-L1 inhibitor naïve participants with received isatuximab 10 mg/kg, IV infusion QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days), and then Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, with optional radiotherapy until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort B: DLBCL: Isatuximab + Cemiplimab: DLBCL, anti PD-1/PD-L1 naïve participants with received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 12 | 17 | 11
Participants
  Hyponatremia: Grade 1 | 8 | 4 | 6 | 5
  Hyponatremia: Grade 2 | 0 | 0 | 0 | 0
  Hyponatremia: Grade 3 | 0 | 0 | 2 | 3
  Hyponatremia: Grade 4 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 1 | 0 | 0 | 0 | 0
  Hypokalemia: Grade 2 | 3 | 3 | 3 | 5
  Hypokalemia: Grade 3 | 0 | 0 | 3 | 0
  Hypokalemia: Grade 4 | 0 | 0 | 0 | 0
  Hyperkalemia: Grade 1 | 1 | 2 | 2 | 1
  Hyperkalemia: Grade 2 | 1 | 0 | 0 | 1
  Hyperkalemia: Grade 3 | 0 | 0 | 0 | 1
  Hyperkalemia: Grade 4 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 1: number analyzed (Participants) | 5 | 6 | 4 | 3
  Hypocalcemia: Grade 1 | 1 | 0 | 1 | 1
  Hypocalcemia: Grade 2: number analyzed (Participants) | 5 | 6 | 4 | 3
  Hypocalcemia: Grade 2 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 3: number analyzed (Participants) | 5 | 6 | 4 | 3
  Hypocalcemia: Grade 3 | 0 | 0 | 0 | 0
  Hypocalcemia: Grade 4: number analyzed (Participants) | 5 | 6 | 4 | 3
  Hypocalcemia: Grade 4 | 0 | 0 | 0 | 0
  Hypoalbuminemia: Grade 1 | 3 | 2 | 5 | 2
  Hypoalbuminemia: Grade 2 | 4 | 0 | 6 | 5
  Hypoalbuminemia: Grade 3 | 0 | 0 | 0 | 1
  Hypoalbuminemia: Grade 4 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 1 | 5 | 1 | 0 | 1
  Hypoglycemia: Grade 2 | 0 | 0 | 0 | 1
  Hypoglycemia: Grade 3 | 0 | 0 | 0 | 0
  Hypoglycemia: Grade 4 | 0 | 0 | 0 | 0
  Hyperglycemia: Grade 1 | 2 | 5 | 1 | 6
  Hyperglycemia: Grade 2 | 2 | 2 | 3 | 2
  Hyperglycemia: Grade 3 | 2 | 0 | 1 | 0
  Hyperglycemia: Grade 4 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 1: number analyzed (Participants) | 5 | 6 | 4 | 3
  Hypercalcemia: Grade 1 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 2: number analyzed (Participants) | 5 | 6 | 4 | 3
  Hypercalcemia: Grade 2 | 0 | 0 | 0 | 0
  Hypercalcemia: Grade 3: number analyzed (Participants) | 5 | 6 | 4 | 3
  Hypercalcemia: Grade 3 | 0 | 0 | 1 | 0
  Hypercalcemia: Grade 4: number analyzed (Participants) | 5 | 6 | 4 | 3
  Hypercalcemia: Grade 4 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Laboratory Abnormalities: Renal Parameters
Description: Abnormal renal parameters assessed were glomerular filtration rate (GFR) by class, creatinine increased and hyperuricemia. GFR by class was assessed in categories:>=90 milliliter per minute per 1.73 meter square (mL/min/1.73m^2) (Normal), >=60 to <90 mL/min/1.73m^2 (Mild), >=30 to <60 mL/min/1.73m^2 (Moderate), >=15 to <30 mL/min/1.73m^2 (Severe), and <15 mL/min/1.73m^2 (End Stage Renal Disease). Abnormal criteria was assessed as per NCI-CTCAE v 5.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: up to 103 weeks)
Population: Analysis was performed on all treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 12 | 17 | 11
Participants
  GFR: >=90 mL/min/1.73m^2 | 7 | 2 | 4 | 1
  GFR: >=60 to <90 mL/min/1.73m^2 | 8 | 8 | 8 | 7
  GFR: >=30 to <60 mL/min/1.73m^2 | 3 | 2 | 4 | 2
  GFR: >=15 to <30 mL/min/1.73m^2 | 0 | 0 | 1 | 1
  GFR: <15 mL/min/1.73m^2 | 0 | 0 | 0 | 0
  Creatinine increased: Grade 1 | 2 | 3 | 4 | 1
  Creatinine increased: Grade 2 | 3 | 1 | 3 | 4
  Creatinine increased: Grade 3 | 0 | 0 | 0 | 0
  Creatinine increased: Garde 4 | 0 | 0 | 0 | 0
  Hyperuricemia: Grade 1 | 0 | 0 | 0 | 0
  Hyperuricemia: Grade 2 | 0 | 0 | 0 | 0
  Hyperuricemia: Grade 3 | 1 | 3 | 5 | 2
  Hyperuricemia: Grade 4 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Laboratory Abnormalities: Liver Function Parameters
Description: Abnormal liver function parameters assessed were aspartate aminotransferase (AST) increased, alanine aminotransferase (ALT) increased, alkaline phosphatase (ALP) increased, blood bilirubin (BB) increased. Abnormal criteria was assessed as per NCI-CTCAE v 5.0, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: up to 103 weeks)
Population: Analysis was performed on all treated population.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 12 | 17 | 11
Participants
  AST increased: Grade 1 | 3 | 2 | 5 | 3
  AST increased: Grade 2 | 0 | 0 | 1 | 0
  AST increased: Grade 3 | 0 | 0 | 0 | 0
  AST increased: Grade 4 | 0 | 0 | 0 | 0
  ALT increased: Grade 1 | 1 | 7 | 6 | 0
  ALT increased: Grade 2 | 0 | 0 | 0 | 0
  ALT increased: Grade 3 | 0 | 0 | 0 | 0
  ALT increased: Grade 4 | 0 | 0 | 0 | 0
  ALP increased: Grade 1 | 3 | 5 | 4 | 5
  ALP increased: Grade 2 | 2 | 0 | 2 | 0
  ALP increased: Grade 3 | 0 | 0 | 0 | 0
  ALP increased: Grade 4 | 0 | 0 | 0 | 0
  BB increased: Grade 1 | 1 | 0 | 1 | 2
  BB increased: Grade 2 | 0 | 0 | 2 | 1
  BB increased: Grade 3 | 0 | 0 | 1 | 0
  BB increased: Grade 4 | 0 | 0 | 0 | 0

7. Primary Outcome: Cohort A1: Percentage of Participants With Complete Response (CR)
Description: Percentage of participants who had a CR as a best overall response (BOR) using the Lugano response criteria (LRC) 2014 (based on PET-CT and CT responses). Per LRC, CR based on PET-CT response was defined as complete metabolic response (MR) in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass, on 5-point scale (5PS), where, 1= no uptake above background; 2 = uptake <=mediastinum; 3 = uptake > mediastinum but <= liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. CR based on CT-response was defined as target nodes/nodal masses of lymph nodes, extralymphatic sites regressed to <=1.5 cm in longest dimension transverse diameter of lesion (LDi); absence of non-measured lesion; organ enlargement regressed to normal; no new lesions; normal bone marrow morphology; if indeterminate, immunohistochemistry negative.
Time Frame: From the date of randomization until disease progression or death or study cut-off date, whichever comes first (maximum duration: up to 103 weeks)
Population: Analysis was performed on all treated population. Data for this outcome measure was not planned to be collected and analyzed for Cohort B and C as pre-specified in protocol.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18
percentage of participants | 27.8

8. Primary Outcome: Cohort A2, B and C: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants who had a CR or partial response (PR) as BOR using LRC, 2014. Per LRC, CR (PET-CT): complete MR in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass; no new lesions and no evidence of FDG-avid disease. CR (CT-response): target nodes/nodal masses of lymph nodes, extralymphatic sites regressed to <=1.5cm LDi; absence of non-measured lesion; organ enlargement regressed to normal; no new lesions; normal bone marrow morphology. PR (PET-CT): partial MR in lymph nodes and extralymphatic sites; no new lesions and residual uptake higher than uptake. PR (Per CT): lymph nodes, extralymphatic sites>=50% decrease in sum of product of perpendicular diameters (SPD), extranodal sites; if lesion is too small to measure on CT,assign5mm*5mm as default; if no longer visible:0*0mm; Node>5mm*5mm but smaller than normal, use actual measurement; absent/regressed non-measured lesions; no increase; spleen regressed by>50% or no new lesions.
Time Frame: From the date of randomization until disease progression, or death or study cut-off date, whichever comes first (maximum duration: up to 103 weeks)
Population: Analysis was performed on all treated population.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cohort C: PTCL: Isatuximab + Cemiplimab: PTCL, anti PD-1/PD-L1 naïve participants with received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 12 | 17 | 11
percentage of participants | 33.3 [12.3 to 60.9] | 5.9 [0.3 to 25.0] | 9.1 [0.5 to 36.4]

9. Secondary Outcome: Number of Participants With Treatment-Induced and Treatment Boosted Antidrug Antibodies (ADA) Against Isatuximab
Description: ADA responses were categorized as treatment boosted ADA and treatment-induced ADA. Treatment boosted ADA was defined as pre-existing ADAs with a significant increase in the ADA titer during the study compared to the Baseline titer. Treatment-induced ADA was defined as ADA that developed at any time during the ADA on-study observation period in participants without pre-existing ADA.
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: up to 103 weeks)
Population: Analysis was performed on Anti-drug antibody (ADA) evaluable population that included all participants who signed informed consent and received at least 1 dose of either isatuximab or cemiplimab, with at least 1 non-missing ADA result after the drug administration. Here, "overall number of participants" analyzed signifies the participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 17 | 12 | 6 | 5
Participants
  Treatment-Induced ADA | 1 | 0 | 0 | 0
  Treatment-Boosted ADA | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment-Induced and Treatment Boosted Antidrug Antibodies (ADA) Against Cemiplimab
Description: as for outcome 9
Time Frame: From first dose of study treatment up to 30 days after last dose of study treatment (maximum duration: up to 103 weeks)
Population: Analysis was performed on ADA evaluable population. Here, "overall number of participants" analyzed signifies the participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 11 | 10 | 6
Participants
  Treatment-Induced ADA | 0 | 0 | 1 | 0
  Treatment-Boosted ADA | 0 | 0 | 0 | 0

11. Secondary Outcome: Pharmacokinetics (PK) Parameter: Plasma Concentration of Isatuximab at End of Infusion (CEOI)
Description: Ceoi is the plasma concentration observed at the end of intravenous infusion of isatuximab.
Time Frame: End of infusion (EOI up to 3 hours) on Day 2 of Cycle 1
Population: Analysis was performed on PK population (for isatuximab) which included participants who signed informed consent and received at least 1 dose of the drug with at least one reportable concentration after the study drug (isatuximab) administration. Here, "overall number of participants" analyzed signifies the participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Groups:
- Cohort A1: cHL: Isatuximab: cHL, PD-1/PD-L1 inhibitor naïve participants received isatuximab 10 mg/kg, IV infusion QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days), and then Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) with optional radiotherapy, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort A2: cHL: Isatuximab: cHL, anti-PD-1/PD-L1 inhibitor progressor participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) with optional radiotherapy until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort B: DLBCL: Isatuximab: DLBCL, anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days), until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort C: PTCL: Isatuximab: PTCL, anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days), until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Isatuximab | Cohort A2: cHL: Isatuximab | Cohort B: DLBCL: Isatuximab | Cohort C: PTCL: Isatuximab
Number analyzed (Participants) | 17 | 12 | 14 | 7
micrograms per milliliter (mcg/mL) | 221 (47.2) | 263 (39.4) | 235 (39.3) | 181 (35.7)

12. Secondary Outcome: PK Parameter: Maximum Observed Plasma Concentration (Cmax) After the First Infusion of Isatuximab
Description: Cmax was defined as the maximum plasma concentration observed after the first administration of drug.
Time Frame: At Start of infusion (SOI; 0 hour), before actual EOI (up to 3 hours), EOI+ 4 hours, 72 hours and 144 hours post-dose on Day 2 of Cycle 1
Population: Analysis was performed on PK population (for isatuximab). Here, "overall number of participants" analyzed signifies the participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort A1: cHL: Isatuximab | Cohort A2: cHL: Isatuximab | Cohort B: DLBCL: Isatuximab | Cohort C: PTCL: Isatuximab
Number analyzed (Participants) | 17 | 12 | 14 | 7
mcg/mL | 226 (48.1) | 265 (38.8) | 253 (29.1) | 181 (35.7)

13. Secondary Outcome: PK Parameter: Time to Reach Cmax (Tmax) After the First Infusion of Isatuximab
Description: Tmax was defined as the time to reach Cmax, after the intravenous infusion of isatuximab.
Time Frame: At SOI (0 hour), before actual EOI (up to 3 hours), EOI+ 4 hours, 72 hours and 144 hours post-dose on Day 2 of Cycle 1
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A1: cHL: Isatuximab | Cohort A2: cHL: Isatuximab | Cohort B: DLBCL: Isatuximab | Cohort C: PTCL: Isatuximab
Number analyzed (Participants) | 17 | 12 | 14 | 7
hours | 5.95 [2.00 to 8.92] | 5.23 [3.00 to 8.83] | 5.26 [2.60 to 10.5] | 4.57 [2.33 to 7.45]

14. Secondary Outcome: PK Parameter: Area Under the Plasma Concentration (AUClast) Versus Time Curve After the First Infusion of Isatuximab
Description: AUClast was defined as area under the plasma concentration versus time curve calculated from time 0 to last quantifiable concentration, calculated for isatuximab.
Time Frame: At SOI (0 hour), before actual EOI (up to 3 hours), EOI+ 4 hours, 72 hours and 144 hours post-dose on Day 2 of Cycle 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours*mcg/mL
Groups:
- Cohort B: DLBCL: Isatuximab: DLBCL, anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Isatuximab | Cohort A2: cHL: Isatuximab | Cohort B: DLBCL: Isatuximab | Cohort C: PTCL: Isatuximab
Number analyzed (Participants) | 17 | 12 | 14 | 7
hours*mcg/mL | 20400 (5190) | 22700 (6020) | 21700 (4610) | 14400 (4710)

15. Secondary Outcome: PK Parameter: Last Concentration Observed Above the Lower Limit of Quantification (Clast) After the First Infusion of Isatuximab
Description: Clast was defined as the last concentration of isatuximab observed above the lower limit of quantification.
Time Frame: At SOI (0 hour), before actual EOI (up to 3 hours), EOI+ 4 hours, 72 hours and 144 hours post-dose on Day 2 of Cycle 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort A1: cHL: Isatuximab | Cohort A2: cHL: Isatuximab | Cohort B: DLBCL: Isatuximab | Cohort C: PTCL: Isatuximab
Number analyzed (Participants) | 17 | 12 | 14 | 7
mcg/mL | 93.3 (28.1) | 110 (24.5) | 89.8 (24.7) | 40.4 (17.7)

16. Secondary Outcome: PK Parameter: Time of Clast (Tlast) After the First Infusion of Isatuximab
Description: Tlast was defined as the time of last concentration observed above the lower limit of quantification for isatuximab.
Time Frame: At SOI (0 hour), before actual EOI (up to 3 hours), EOI+ 4 hours, 72 hours and 144 hours post-dose on Day 2 of Cycle 1
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A1: cHL: Isatuximab | Cohort A2: cHL: Isatuximab | Cohort B: DLBCL: Isatuximab | Cohort C: PTCL: Isatuximab
Number analyzed (Participants) | 17 | 12 | 14 | 7
hours | 142 [136 to 174] | 143 [72.6 to 167] | 143 [137 to 147] | 144 [142 to 169]

17. Secondary Outcome: PK Parameter: Area Under the Concentration Versus Time Curve Over the Dosing Interval (AUC0-168 Hours) After the First Infusion of Isatuximab
Description: AUC0-168 hours was defined as the area under the plasma concentration versus time curve from time 0 to 168 hours post dose calculated for isatuximab. Samples for this outcome measure were collected up to 144 hours post-dose. No sample was collected at 168 hours post-dose; and thus, the samples collected up to 144 hours post-dose were extrapolated to derive data for 168 hours post-dose.
Time Frame: At SOI (0 hour), before actual EOI (up to 3 hours), EOI+ 4 hours, 72 hours and 144 hours post-dose on Day 2 of Cycle 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hour*mcg/mL
Arm/Group | Cohort A1: cHL: Isatuximab | Cohort A2: cHL: Isatuximab | Cohort B: DLBCL: Isatuximab | Cohort C: PTCL: Isatuximab
Number analyzed (Participants) | 17 | 11 | 14 | 7
hour*mcg/mL | 22500 (5770) | 26600 (4030) | 23700 (4960) | 15000 (4680)

18. Secondary Outcome: PK Parameter: Area Under the Concentration Versus Time Curve Over the Dosing Interval (AUC0-144 Hours) After the First Infusion of Isatuximab
Description: AUC0-144 hours was defined as the area under the plasma concentration versus time curve from time 0 to 144 hours post dose calculated for isatuximab.
Time Frame: At SOI (0 hour), before actual EOI (up to 3 hours), EOI+ 4 hours, 72 hours and 144 hours post-dose on Day 2 of Cycle 1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours*mcg/mL
Arm/Group | Cohort A1: cHL: Isatuximab | Cohort A2: cHL: Isatuximab | Cohort B: DLBCL: Isatuximab | Cohort C: PTCL: Isatuximab
Number analyzed (Participants) | 17 | 11 | 14 | 7
hours*mcg/mL | 20400 (5170) | 24300 (3470) | 21800 (4550) | 14000 (4240)

19. Secondary Outcome: PK Parameter: Plasma Trough Concentration (Ctrough) of Isatuximab
Description: Ctrough was the plasma concentration of isatuximab observed just before treatment administration during repeated dosing.
Time Frame: Pre-infusion on Cycle1:Day 2, 8, 15, & 22, Cycle 2:Day 1 &15, Cycle 3:Day 1 &15, Cycle 4:Day 1 &15, Cycle 5 Day1,Cycle 6 Day1,Cycle 7 Day 1, Cycle 8 Day1, Cycle 9 Day1, Cycle 10 Day1, Cycle 11 Day1, Cycle14 Day1, Cycle 17 Day1, Cycle 20 Day1,Cycle 23 Day1
Population: Analysis was performed on PK population (for isatuximab). Here, '0' in the number analyzed field signifies that none of the participants were available for the specified timepoints.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort A1: cHL: Isatuximab | Cohort A2: cHL: Isatuximab | Cohort B: DLBCL: Isatuximab | Cohort C: PTCL: Isatuximab
Number analyzed (Participants) | 18 | 12 | 16 | 9
mcg/mL
  Cycle 1 Day 2: number analyzed (Participants) | 18 | 12 | 15 | 9
  Cycle 1 Day 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Cycle 1 Day 8: number analyzed (Participants) | 17 | 10 | 15 | 8
  Cycle 1 Day 8 | 93.1 (28.1) | 98.4 (39.5) | 93.2 (27.2) | 37.7 (18.0)
  Cycle 1 Day 15: number analyzed (Participants) | 16 | 8 | 10 | 6
  Cycle 1 Day 15 | 159 (47.7) | 191 (41.4) | 181 (43.7) | 115 (89.4)
  Cycle 1 Day 22: number analyzed (Participants) | 13 | 12 | 9 | 5
  Cycle 1 Day 22 | 254 (59.8) | 262 (45.2) | 259 (57.9) | 124 (22.9)
  Cycle 2 Day 1: number analyzed (Participants) | 15 | 9 | 5 | 4
  Cycle 2 Day 1 | 310 (78.2) | 352 (48.7) | 316 (110) | 132 (64.0)
  Cycle 2 Day 15: number analyzed (Participants) | 15 | 10 | 5 | 5
  Cycle 2 Day 15 | 314 (141) | 390 (256) | 291 (108) | 129 (59.1)
  Cycle 3 Day 1: number analyzed (Participants) | 17 | 10 | 5 | 5
  Cycle 3 Day 1 | 304 (79.8) | 320 (49.7) | 327 (92.4) | 122 (58.0)
  Cycle 3 Day 15: number analyzed (Participants) | 15 | 11 | 3 | 3
  Cycle 3 Day 15 | 325 (85.1) | 336 (42.3) | 420 (67.8) | 176 (8.19)
  Cycle 4 Day 1: number analyzed (Participants) | 14 | 11 | 2 | 4
  Cycle 4 Day 1 | 334 (91.8) | 344 (58.2) | 350 (80.6) | 149 (33.2)
  Cycle 4 Day 15: number analyzed (Participants) | 15 | 9 | 2 | 3
  Cycle 4 Day 15 | 363 (122) | 376 (65.2) | 336 (117) | 158 (16.9)
  Cycle 5 Day 1: number analyzed (Participants) | 13 | 10 | 1 | 3
  Cycle 5 Day 1 | 385 (79.9) | 383 (71.0) | 362 | 157 (11.5)
  Cycle 6 Day 1: number analyzed (Participants) | 11 | 7 | 1 | 1
  Cycle 6 Day 1 | 379 (105) | 361 (97.8) | 415 | 137
  Cycle 7 Day 1: number analyzed (Participants) | 9 | 8 | 0 | 1
  Cycle 7 Day 1 | 408 (141) | 374 (107) |  | 186
  Cycle 8 Day 1: number analyzed (Participants) | 9 | 6 | 1 | 0
  Cycle 8 Day 1 | 352 (94.9) | 356 (57.7) | 360 |
  Cycle 9 Day 1: number analyzed (Participants) | 8 | 6 | 0 | 1
  Cycle 9 Day 1 | 328 (124) | 351 (54.8) |  | 83.5
  Cycle 10 Day 1: number analyzed (Participants) | 7 | 5 | 1 | 0
  Cycle 10 Day 1 | 317 (120) | 347 (51.8) | 383 |
  Cycle 11 Day 1: number analyzed (Participants) | 5 | 5 | 0 | 0
  Cycle 11 Day 1 | 318 (147) | 357 (52.0) |  |
  Cycle 14 Day 1: number analyzed (Participants) | 3 | 5 | 0 | 0
  Cycle 14 Day 1 | 357 (119) | 333 (28.0) |  |
  Cycle 17 Day 1: number analyzed (Participants) | 0 | 5 | 0 | 0
  Cycle 17 Day 1 |  | 299 (22.3) |  |
  Cycle 20 Day 1: number analyzed (Participants) | 1 | 4 | 0 | 0
  Cycle 20 Day 1 | 117 | 328 (14.4) |  |
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 2 | 0 | 0
  Cycle 23 Day 1 |  | 309 (9.90) |  |

20. Secondary Outcome: PK Parameter: Serum Concentration of Cemiplimab at End of Infusion (CEOI)
Description: Ceoi is the plasma concentration observed at the end of intravenous infusion of cemiplimab.
Time Frame: EOI (up to 30 minutes [min]) on Day 1 of Cycle 1
Population: Analysis was performed on PK population (for Cemiplimab) which included all participants who signed informed consent and received at least 1 dose of the drug with at least one reportable concentration after the study drug (cemiplimab) administration. Here 'overall number of participants analyzed" signifies the participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams per milliliter (mg/mL)
Groups:
- Cohort A1: cHL: Cemiplimab: cHL, PD-1/PD-L1 inhibitor naïve participants received cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 (each cycle of 28 days) and then 350 mg Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days), with optional radiotherapy until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort A2: cHL: Cemiplimab: cHL, anti-PD-1/PD-L1 inhibitor progressor participants received cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 (each cycle of 28 days) and then 350 mg Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days), with optional radiotherapy until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort B: DLBCL: Cemiplimab: DLBCL, anti PD-1/PD-L1 naïve participants received cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort C: PTCL: Cemiplimab: PTCL, anti PD-1/PD-L1 naïve participants received cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 (each cycle of 28 days) and then 350 mg Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Cemiplimab | Cohort A2: cHL: Cemiplimab | Cohort B: DLBCL: Cemiplimab | Cohort C: PTCL: Cemiplimab
Number analyzed (Participants) | 17 | 5 | 15 | 8
milligrams per milliliter (mg/mL) | 63.7 (24.2) | 78.8 (24.9) | 68.1 (26.3) | 66.2 (18.4)

21. Secondary Outcome: PK Parameter: Maximum Observed Concentration (Cmax) After the First Infusion of Cemiplimab
Description: Cmax was defined as the maximum concentration observed after the first administration.
Time Frame: At SOI (0 hour), before actual EOI (up to 30 min), EOI+4 hours, 96 hours, 168 hours, and 336 hours post-dose on Day 1 of Cycle 1
Population: Analysis was performed on PK population (for Cemiplimab). Here, "overall number of participants" analyzed signifies the participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Cohort B: DLBCL: Cemiplimab: DLBCL, anti PD-1/PD-L1 naïve participants received cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 (each cycle of 28 days) and then 350 mg Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days), until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort C: PTCL: Cemiplimab: PTCL, anti PD-1/PD-L1 naïve participants received cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 (each cycle of 28 days) and then 350 mg Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days), until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Cemiplimab | Cohort A2: cHL: Cemiplimab | Cohort B: DLBCL: Cemiplimab | Cohort C: PTCL: Cemiplimab
Number analyzed (Participants) | 17 | 5 | 15 | 8
mg/L | 70.9 (21.1) | 90.8 (19.4) | 79.0 (16.7) | 77.1 (20.7)

22. Secondary Outcome: PK Parameter: Time to Reach Cmax (Tmax) After the First Infusion of Cemiplimab
Description: Tmax was defined as the time to reach Cmax after the intravenous infusion of cemiplimab.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Median (Full Range); unit: hours
Groups:
- Cohort B: DLBCL: Cemiplimab: DLBCL, anti PD-1/PD-L1 naïve participants received cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 (each cycle of 28 days) and then 350 mg Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Cemiplimab | Cohort A2: cHL: Cemiplimab | Cohort B: DLBCL: Cemiplimab | Cohort C: PTCL: Cemiplimab
Number analyzed (Participants) | 17 | 5 | 15 | 8
hours | 4.00 [0.480 to 4.67] | 4.50 [0.480 to 4.53] | 4.05 [0.420 to 5.40] | 2.34 [0.500 to 4.08]

23. Secondary Outcome: PK Parameter: Area Under the Serum Concentration (AUClast) Versus Time Curve After the First Infusion of Cemiplimab
Description: AUClast was defined as area under the serum concentration versus time curve calculated from time 0 to last quantifiable concentration calculated for cemiplimab.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: day*mg/mL
Groups:
- Cohort C: PTCL: Isatuximab + Cemiplimab: PTCL, anti PD-1/PD-L1 naïve participants received cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 (each cycle of 28 days) and then 350 mg Q3W from Cycle 7 to Cycle 30 (each cycle of 28 days) until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Cemiplimab | Cohort A2: cHL: Cemiplimab | Cohort B: DLBCL: Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 17 | 5 | 15 | 8
day*mg/mL | 524 (188) | 648 (112) | 506 (159) | 466 (147)

24. Secondary Outcome: PK Parameter: Last Concentration Observed Above the Lower Limit of Quantification (Clast) After the First Infusion of Cemiplimab
Description: Clast was defined as the last concentration of cemiplimab observed above the lower limit of quantification.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cohort A1: cHL: Cemiplimab | Cohort A2: cHL: Cemiplimab | Cohort B: DLBCL: Cemiplimab | Cohort C: PTCL: Cemiplimab
Number analyzed (Participants) | 17 | 5 | 15 | 8
mg/L | 23.4 (11.2) | 30.3 (7.16) | 27.0 (9.79) | 14.3 (6.64)

25. Secondary Outcome: PK Parameter: Time of Clast (Tlast) After the First Infusion of Cemiplimab
Description: Tlast was defined as the time of last concentration observed above the lower limit of quantification for cemiplimab.
Time Frame: as for outcome 21
Population: Analysis was performed on PK population (for Cemiplimab). Here, "overall number of participants analyzed" signifies the participants with available data for this outcome measure.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort A1: cHL: Cemiplimab | Cohort A2: cHL: Cemiplimab | Cohort B: DLBCL: Cemiplimab | Cohort C: PTCL: Cemiplimab
Number analyzed (Participants) | 17 | 5 | 15 | 8
hours | 334 [164 to 672] | 333 [330 to 362] | 332 [164 to 339] | 335 [171 to 572]

26. Secondary Outcome: PK Parameter: Area Under the Serum Concentration Versus Time Curve Over the Dosing Interval (AUC0-336 Hours) After the First Infusion of Cemiplimab
Description: AUC0-336 hours was defined as the area under the serum concentration versus time curve from time 0 to 336 hours post dose for cemiplimab.
Time Frame: as for outcome 21
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: day*mg/mL
Arm/Group | Cohort A1: cHL: Cemiplimab | Cohort A2: cHL: Cemiplimab | Cohort B: DLBCL: Cemiplimab | Cohort C: PTCL: Cemiplimab
Number analyzed (Participants) | 17 | 5 | 15 | 8
day*mg/mL | 519 (177) | 645 (113) | 546 (136) | 466 (130)

27. Secondary Outcome: PK Parameter: Serum Trough Concentration (Ctrough) of Cemiplimab
Description: Ctrough was the serum concentration of cemiplimab observed just before treatment administration during repeated dosing.
Time Frame: Pre-infusion on Cycle 1:Day 1 & Day15,Cycle 2:Day 1 & Day 15,Cycle 3:Day 1 & Day 15,Cycle 4:Day 1 & Day15,Cycle 5 Day 1,Cycle 6 Day 1,Cycle7 Day1,Cycle 8 Day 1,Cycle 9 Day1,Cycle 10 Day1,Cycle11 Day1,Cycle14 Day 1,Cycle 17 Day1,Cycle20 Day 1,Cycle 23 Day1
Population: Analysis was performed on PK population (for Cemiplimab). Here, '0' in the number analyzed field signifies that none of the participants were available for the specified timepoint.
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Cohort A1: cHL: Cemiplimab | Cohort A2: cHL: Cemiplimab | Cohort B: DLBCL: Cemiplimab | Cohort C: PTCL: Cemiplimab
Number analyzed (Participants) | 18 | 12 | 17 | 11
mg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 17 | 5 | 17 | 11
  Cycle 1 Day 1 | 0.00800 (0.0330) | 0.980 (2.19) | 0 (0) | 0 (0)
  Cycle 1 Day 15: number analyzed (Participants) | 14 | 5 | 12 | 6
  Cycle 1 Day 15 | 25.3 (10.2) | 30.3 (7.16) | 24.2 (9.91) | 16.5 (4.83)
  Cycle 2 Day 1: number analyzed (Participants) | 14 | 5 | 5 | 4
  Cycle 2 Day 1 | 44.1 (11.2) | 51.1 (15.8) | 49.6 (16.3) | 33.0 (10.4)
  Cycle 2 Day 15: number analyzed (Participants) | 14 | 4 | 5 | 5
  Cycle 2 Day 15 | 64.4 (22.5) | 61.0 (10.8) | 48.9 (9.16) | 38.3 (21.1)
  Cycle 3 Day 1: number analyzed (Participants) | 16 | 5 | 5 | 5
  Cycle 3 Day 1 | 77.7 (30.2) | 73.7 (11.0) | 62.8 (13.6) | 66.7 (64.7)
  Cycle 3 Day 15: number analyzed (Participants) | 13 | 5 | 3 | 3
  Cycle 3 Day 15 | 95.1 (35.0) | 86.6 (19.5) | 72.3 (3.80) | 72.1 (12.1)
  Cycle 4 Day 1: number analyzed (Participants) | 13 | 5 | 2 | 4
  Cycle 4 Day 1 | 100 (38.9) | 84.4 (20.3) | 76.8 (4.31) | 66.7 (24.1)
  Cycle 4 Day 15: number analyzed (Participants) | 13 | 4 | 2 | 3
  Cycle 4 Day 15 | 113 (44.8) | 88.2 (30.5) | 91.6 (10.3) | 63.5 (24.8)
  Cycle 5 Day 1: number analyzed (Participants) | 12 | 4 | 1 | 3
  Cycle 5 Day 1 | 106 (28.9) | 92.7 (21.8) | 91.6 | 73.4 (26.5)
  Cycle 6 Day 1: number analyzed (Participants) | 10 | 4 | 1 | 1
  Cycle 6 Day 1 | 114 (37.3) | 94.8 (29.8) | 113 | 73.8
  Cycle 7 Day 1: number analyzed (Participants) | 8 | 5 | 0 | 1
  Cycle 7 Day 1 | 112 (32.6) | 115 (43.0) |  | 100
  Cycle 8 Day 1: number analyzed (Participants) | 9 | 3 | 1 | 0
  Cycle 8 Day 1 | 110 (40.5) | 129 (19.5) | 93.0 |
  Cycle 9 Day 1: number analyzed (Participants) | 7 | 3 | 1 | 1
  Cycle 9 Day 1 | 107 (36.2) | 122 (27.9) | 122 | 61.8
  Cycle 10 Day 1: number analyzed (Participants) | 7 | 3 | 1 | 0
  Cycle 10 Day 1 | 112 (65.8) | 139 (23.2) | 122 |
  Cycle 11 Day 1: number analyzed (Participants) | 6 | 4 | 0 | 0
  Cycle 11 Day 1 | 120 (60.2) | 133 (14.5) |  |
  Cycle 14 Day 1: number analyzed (Participants) | 3 | 4 | 0 | 0
  Cycle 14 Day 1 | 138 (72.7) | 127 (17.1) |  |
  Cycle 17 Day 1: number analyzed (Participants) | 1 | 4 | 0 | 0
  Cycle 17 Day 1 | 60.6 | 131 (18.8) |  |
  Cycle 20 Day 1: number analyzed (Participants) | 1 | 3 | 0 | 0
  Cycle 20 Day 1 | 62.6 | 137 (26.7) |  |
  Cycle 23 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 0
  Cycle 23 Day 1 |  | 137 |  |

28. Secondary Outcome: Percent Change From Baseline in Tumor Burden
Description: Tumor burden change was defined as the best percent-change from baseline in a sum of product of lesion diameters (longest for non-nodal lesion, short axis for nodal lesions) for all target lesions.
Time Frame: Up to 103 weeks
Population: Analysis was performed on all treated population. Here, "overall number of participants" analyzed signifies the participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Cohort A1: cHL: Isatuximab + Cemiplimab: cHL, PD-1/PD-L1 inhibitor naïve participants received isatuximab 10 mg/kg, IV infusion QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days), and then Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, with optional radiotherapy, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 10 | 8 | 6
percent change | -48.8 (59.0) | -55.3 (32.6) | 396.0 (880.7) | -9.7 (87.8)

29. Secondary Outcome: Duration of Response (DOR)
Description: Time (months) between date of first response to first date that recurrent or radiologically disease progression (PD) was documented, or date of death,whichever was 1st. In absence of PD or death before cut-off date or date of initiation of further anticancer treatment, DOR was censored at date of last valid response not showing PD performed prior to initiation of further anticancer treatment or cut-off date, whichever was earlier. PD(PET-CT): metabolic disease with score 4/5 with inc. in intensity of uptake for target nodes/nodal mass & new FDG-avid foci consistent with lymphoma. PD(CT):any 1 of following: cross product of longest transverse diameter of lesion(LDi) & perpendicular diameter (PPD) progression of nodes/nodal mass, abnormal node/lesion with LDi >1.5 cm, inc >=50% from PPD nadir & inc in LDi/ shortest axis perpendicular to LDi(SDi) from nadir 0.5 cm, regrowth of resolved lesions, new splenomegaly,progression of non-measured lesion, new/recurrent involvement of bone marrow.
Time Frame: From the date of first response until disease progression or death, or study cut-off date whichever occurred first (maximum duration: up to 103 weeks)
Population: Analysis was performed on participants who had a response. DOR was analyzed using Kaplan-Meier method. Here, "overall number of participants" analyzed signifies the participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 10 | 4 | 1 | 1
months | 5.8 (5.2) | 7.3 (4.8) | 17.1 | 14.0

30. Secondary Outcome: Percentage of Participants With Disease Control (DC)
Description: DC defined as percentage of participants who achieved CR, PR or stable disease (SD) as per LRC, 2014. CR (PET-CT): complete MR in lymph nodes and extralymphatic sites; no new lesions and no evidence of FDG-avid disease. CR (CT): target nodes/nodal masses of lymph nodes, extralymphatic sites regressed to <=1.5cm LDi; absence of non-measured lesion; organ enlargement regressed to normal; no new lesions; normal bone marrow. PR (PET-CT): partial MR in lymph nodes and sites; no new lesions. PR (CT): lymph nodes, sites>=50% decrease in SPD, sites; if lesion is too small to measure on CT, assign 5mm*5mm; No longer visible:0*0mm; Node>5mm*5mm, use actual measurement; absent/regressed non-measured lesions; no increase; spleen regressed by>50% or no new lesions. SD (PET-CT):no metabolic response, target nodes score of 4/5 with no significant change & no new lesions; SD (CT): <50% dec in SPD, no increase in progression for. 5PS:1: non-measured lesions, organ enlargement & no new lesions.
Time Frame: as for outcome 29
Population: Analysis was performed on all treated population.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cohort A1: cHL: Isatuximab + Cemiplimab: cHL, PD-1/PD-L1 inhibitor naïve participants received isatuximab 10 mg/kg, IV infusion QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days), and then Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion Q2W from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, with optional radiotherapy, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort A2: cHL: Isatuximab + Cemiplimab: cHL, anti-PD-1/PD-L1 inhibitor progressor participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion Q2W from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, with optional radiotherapy until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort B: DLBCL: Isatuximab + Cemiplimab: DLBCL, anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion Q2W from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
- Cohort C: PTCL: Isatuximab + Cemiplimab: PTCL, anti PD-1/PD-L1 naïve participants received isatuximab 10 mg/kg, IV infusion, QW in Cycle 1 and then Q2W from Cycle 2 to Cycle 6 (each cycle of 28 days) and Q3W from Cycle 7 to Cycle 30 (each cycle of 21 days) along with cemiplimab 250 mg Q2W, IV infusion Q2W from Cycle 1 to 6 and then 350 mg Q3W from Cycle 7 to Cycle 30, until unacceptable AEs or participant's decision to stop the treatment, or at least 96 weeks (at least 48 weeks from initial signal of CR, whichever was longer) of delivery of investigational medicinal product(s) without documented PD, or study cut-off date, whichever occurs first (maximum duration: up to 103 weeks).
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 12 | 17 | 11
percentage of participants | 61.1 [39.2 to 80.1] | 58.3 [31.5 to 81.9] | 5.9 [0.3 to 25.0] | 18.2 [3.3 to 47.0]

31. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS: time (in months) from 1st study treatment administration to date of 1st documented radiographic progression or date of death from any cause, whichever occurs 1st. Per LRC, 2014 PD (per PET-CT): metabolic disease with score 4/5 with increase (inc) in intensity of uptake for individual target nodes/nodal mass & new FDG-avid foci consistent with lymphoma at interim/ end-of-treatment assessment for extra nodal lesions, new FDG-avid foci consistent with lymphoma rather; new/recurrent FDG-avid foci bone marrow. PD (per CT response): any 1 of following: cross product of longest transverse diameter of lesion (LDi) & perpendicular diameter (PPD) progression of nodes/nodal mass, abnormal node/lesion with LDi >1.5 cm, inc >=50% from PPD nadir & inc in LDi/ shortest axis perpendicular to LDi from nadir 0.5 cm for lesion <= 2 cm, regrowth of resolved lesions, new splenomegaly,progression of preexisting non measured lesion, new/recurrent involvement of bone marrow.
Time Frame: as for outcome 8
Population: Analysis was performed on all treated population. PFS was analyzed using Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 12 | 17 | 11
months | 5.09 [2.694 to 13.207] | 6.21 [2.595 to 10.349] | 2.37 [0.460 to 2.694] | 2.66 [0.427 to 6.341]

32. Secondary Outcome: Cohort A1 and A2: Percentage of Participants With Objective Response
Description: Percentage of participants who had a CR or PR as BOR using LRC, 2014 (based on PET-CT and CT responses). CR (per PET-CT): complete MR in lymph nodes and extra lymphatic sites with a score of 1, 2, or 3 with or without residual mass; no new lesions and no evidence of FDG-avid disease. CR (CT-response): target nodes/nodal masses of lymph nodes, extralymphatic sites regressed to <=1.5cm LDi; absence of non-measured lesion; organ enlargement regressed to normal; no new lesions; normal bone marrow morphology. PR (per PET-CT): partial MR in lymph nodes and extral ymphatic sites; no new lesions and residual uptake higher than uptake. PR (per CT): lymph nodes, extralymphatic sites >=50% decrease in SPD, extranodal sites; if lesion is too small to measure on CT, assign 5mm*5mm as default; if no longer visible:0*0mm; Node>5mm*5mm but smaller than normal, used actual measurement; absent/regressed non-measured lesions; no increase; spleen regressed by>50% or no new lesions.
Time Frame: as for outcome 8
Population: Analysis was performed on all treated population. Data for cohort B and C are reported separately.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 12
percentage of participants | 55.6 [34.1 to 75.6] | 33.3 [12.3 to 60.9]

33. Secondary Outcome: Cohort A1 and A2: Percentage of Participants With Complete Response
Description: Percentage of participants who had a CR as a BOR using the LRC, 2014 (based on PET-CT and CT responses). Per LRC, CR based on PET-CT was defined as complete MR in lymph nodes and extralymphatic sites with a score of 1, 2, or 3 with or without residual mass, on 5PS, where, 1= no uptake above background; 2 = uptake <=mediastinum; 3 = uptake > mediastinum but <= liver; 4 = uptake moderately > liver; 5 = uptake markedly higher than liver and/or new lesions; no new lesions and no evidence of FDG-avid disease in bone marrow. CR based on CT-response was defined as target nodes/nodal masses of lymph nodes, extralymphatic sites regressed to <=1.5 cm in longest dimension transverse diameter of lesion (LDi); absence of non-measured lesion; organ enlargement regressed to normal; no new lesions; normal bone marrow morphology; if indeterminate, immunohistochemistry negative.
Time Frame: as for outcome 8
Population: Analysis was performed on all treated population. Data for this outcome measure was not planned to be collected and analyzed for Cohort B and C as pre-specified.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab
Number analyzed (Participants) | 18 | 12
percentage of participants | 27.8 | 16.7

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug (maximum duration: up to 103 weeks)
Description: Analysis was performed on all-treated population.
Arm/Group | Cohort A1: cHL: Isatuximab + Cemiplimab | Cohort A2: cHL: Isatuximab + Cemiplimab | Cohort B: DLBCL: Isatuximab + Cemiplimab | Cohort C: PTCL: Isatuximab + Cemiplimab
All-Cause Mortality (participants affected / at risk) | 4/18 | 0/12 | 12/17 | 6/11
Serious Adverse Events (participants affected / at risk) | 3/18 | 2/12 | 10/17 | 7/11
Other Adverse Events (participants affected / at risk) | 16/18 | 12/12 | 17/17 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1: cHL: Isatuximab + Cemiplimab (N=18) | Cohort A2: cHL: Isatuximab + Cemiplimab (N=12) | Cohort B: DLBCL: Isatuximab + Cemiplimab (N=17) | Cohort C: PTCL: Isatuximab + Cemiplimab (N=11)
Epstein-Barr Virus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster Disseminated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis Aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Haemophilus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Respiratory Syncytial Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Sensorimotor Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual Acuity Reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subclavian Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Performance Status Decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1: cHL: Isatuximab + Cemiplimab (N=18) | Cohort A2: cHL: Isatuximab + Cemiplimab (N=12) | Cohort B: DLBCL: Isatuximab + Cemiplimab (N=17) | Cohort C: PTCL: Isatuximab + Cemiplimab (N=11)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial Diarrhoea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Genital Herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia Staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Stenotrophomonas Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea Cruris (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trichophytosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 3 (6) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vascular Device Infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 2 (2) | 0 (0) | 1 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival Oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear Pruritus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal Discharge Discolouration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0)
Aphthous Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 4 (4) | 4 (6) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epigastric Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 4 (5) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Granulomatous Liver Disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Butterfly Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Milia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash Macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Rash Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1) | 2 (2) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Muscle Tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic Cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration Site Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (4) | 0 (0) | 3 (3) | 1 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 4 (5) | 2 (2)
Generalised Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 3 (3) | 0 (0) | 5 (5) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (7) | 3 (3) | 3 (3) | 3 (3)
Swelling Face (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gamma-Glutamyltransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight Decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Weight Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 7 (11) | 9 (17) | 8 (8) | 7 (8)
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The efficacy results observed in Cohorts B and C did not fulfill the pre-planned interim analysis criteria allowing the study to move to Phase 2 Stage 2 in these cohorts. The efficacy results observed in Cohort A1 and A2 fulfilled the pre-planned interim analysis criteria in Stage 1 to move to Phase 2 Stage 2 in these cohorts. However, the study was stopped for all the cohorts as per Sponsor's decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT03769181/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT03769181/SAP_001.pdf